CLINICAL TRIAL: NCT03266640
Title: A Pilot Study in the Treatment of Refractory Cytomegalovirus (CMV) Infections With Related Donor CMV Specific Cytotoxic T-cells (CTLs) in Children, Adolescents and Young Adult Recipients
Brief Title: Virus Specific Cytotoxic T-Lymphocytes (CTLs) for Refractory Cytomegalovirus (CMV)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Nationwide Children's Hospital (Other); Johns Hopkins University (Other); University of California, San Francisco (Other); Washington University School of Medicine (Other); Indiana University (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 580; FD006363 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cytomegalovirus Infections; Primary Immune Deficiency Disorder
Keywords: Cytomegalovirus; CMV; cytotoxic t-lymphocytes
MeSH Terms: conditions — Cytomegalovirus Infections; Primary Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: All eligible patients will be given CMV specific CTLs and dose is based on donor source: HLA matched and HLA mismatced
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Refractory CMV (Experimental): Patients with refractory CMV will be given one dose of CMV specific CTLs. HLA matched donors will get Dose 2.5 × 10(4) CD3/kg recipient weight; HLA mismatched will get 0.5x10(4) CD3/kg recipient weight. Additional doses may be given for a total of 5 doses if patients do not have a response to the first dose with a reduction in viral load to normal limits.
  Interventions: Drug: viral specific cytotoxic t-lymphocytes

INTERVENTIONS:
Drug: viral specific cytotoxic t-lymphocytes — CMV specific CTLs will be collected from HLA matched or mismatched donors and manufactured in a GMP facility and administered to patients with refractory CMV infection.
  Other Names: CMV CTLs

SUMMARY:
CMV cytotoxic T cells (CTLs) manufactured with the Miltenyi CliniMACS Prodigy Cytokine Capture System will be administered in children, adolescents and young adults (CAYA) with refractory cytomegalovirus (CMV) infection post Allogeneic Hematopoietic Stem Cell Transplantation (AlloHSCT), with primary immunodeficiencies (PID) or post solid organ transplant.

Funding Source: FDA OOPD

ELIGIBILITY:
1. Patients with refractory CMV infection post allogeneic HSCT, with primary immunodeficiencies or post solid organ transplant with either

* Increasing or persistent quantitative qRT-PCR DNA copies despite two weeks of appropriate anti-viral therapy AND/OR
* Medical intolerance to anti-viral therapies including:
* ANC < 500/mm2 secondary to ganciclovir

  * 2 renal toxicity with foscarnet And/or
* known resistance to ganciclovir and/or foscarnet

Consent: Written informed consent given (by patient or legal representative) prior to any study-related procedures.

Performance Status > 30% (Lansky < 16 yrs and Karnofsky > 16 yrs) Age: 0.1 to 79.99 years Females of childbearing potential with a negative urine pregnancy test

Donor Eligibility Related donor available with a T-cell response to the CMV MACS® GMP PepTivator antigen(s).

a. Third Party Allogeneic Donor: If original donor is not available or does not have a T-cell response: third party related allogeneic donor (family donor > 1 HLA A, B, DR match to recipient) with IgG positive to CMV and/or a T-cell response to the CMV MACS® GMP PepTivator .

AND Allogeneic donor disease screening is complete similar to hematopoietic stem cell donors (Appendix 1).

AND Obtained informed consents by donor or donor legally authorized representative prior to donor collection.

3 Patient exclusion criteria:

A patient meeting any of the following criteria is not eligible for the present study:

Patient with acute GVHD > grade 2 or extensive chronic GVHD at the time of CMV CTL infusion Patient receiving steroids (>0.5 mg/kg prednisone equivalent) at the time of CMV CTL infusion Patient treated with donor lymphocyte infusion (DLI) within 4 weeks prior to CMV CTL infusion Thymoglobulin (ATG), Alemtuzumab or T cell immunosuppressive monoclonal antibodies within 30 days Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30% CMV retinitis Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory CMV infection.

Any medical condition which could compromise participation in the study according to the investigator's assessment Known HIV infection Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment.

Known hypersensitivity to iron dextran Patients unwilling or unable to comply with the protocol or unable to give informed consent.

Known human anti-mouse antibodies CMV retinitis, meningitis, encephalitis, and/or cerebritis

Ages: 1 Month to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Patients will be followed for 12 weeks after each infusion
  Patients will be monitored for adverse events following the administration of CMV CTLs
Incidence of Response to Treatment | Patients will be followed 12 weeks after each infusion
  Patients will be followed for improvement in viral infection by monitoring CMV PCR weekly for response to treatment with CTLs

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (9):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided